CLINICAL TRIAL: NCT07081451
Title: The Effect of Guided ımagery Supported Psychoeducation Applied to ındividuals Diagnosed With Depression on Depression, Self-esteem and Stress Level
Acronym: Depression
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kilis 7 Aralik University (Other)
Responsible Party: Principal Investigator, Çiğdem Özdemir, LECTURER, Kilis 7 Aralik University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E.50484
Record Dates: First submitted 2025-05-29; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Depression
Keywords: depression, stress, self-esteem, guided imagery
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group consisting of individuals diagnosed with depression (Experimental): Included 30 patients diagnosed with depression
  Interventions: Other: Guided ımagery supported psychoeducation
- Control group (No Intervention): Included 30 patients diagnosed with depression

INTERVENTIONS:
Other: Guided ımagery supported psychoeducation — Guided Imagery Technique is an effective, economical and therapeutic technique that can be easily used in nursing practices. Guided Imagery Technique is a set of stories that individuals create by visualising the symbols given by the practitioner after relaxation exercises. Within the scope of this technique, which is a window to the inner world of the person, the creation of his/her own unique story through symbols is encouraged
  Other Names: Imagery supported psychoeducation; Guided imagination supported psychoeducation
  Arms: Experimental group consisting of individuals diagnosed with depression

SUMMARY:
Depressive disorder is a common mental disorder. Depression, whose classic symptoms include depressed mood, anxiety, anhedonia and cognitive impairments that profoundly affect quality of life, is one of the leading causes of disability worldwide and the main cause of death by suicide. 3.8% of the world's population suffers from depression, including 5% of adults (4% of men and 6% of women) and 5.7% of those over 60 years of age. Approximately 280 million people worldwide are known to suffer from depression. Depression is often referred to as a stress-related disorder and stress caused by adverse life events, including early in life, is known to contribute to the onset, development and progression of this disorder. Studies have shown that high levels of exposure to negative stressors contribute significantly to cases of depression and that it is important to recognize stress exposures in a timely manner in these individuals. Research has also revealed that self-esteem plays an important role in depression. Self-esteem is defined as "a particular attitude and perception of one's self" that influences one's interactions and feelings towards oneself and others. Low self-esteem has been empirically shown to be a risk factor for the development of depression and suicidal ideation. Low self-esteem is a symptom of depressive disorders and is considered by some to be a precursor to relapse, while high self-esteem seems to buffer against depression. Although effective treatments for depression are available, not all patients receive treatment and of those who do, a significant proportion do not recover. New low-cost and easily accessible ways of dealing with the health burden of depression are increasingly recognized as important. There are a wide range of psychological interventions to treat depression, and one that has been shown to be effective in treating depression is psychoeducation. Psychoeducation is offered to help people with mental disorders understand and manage their illness. It is done by strengthening patients' resources and skills so that they can better cope with their condition, prevent relapse and contribute to their own health and well-being. Studies have shown that psychoeducation programs have positive effects on depression. Another method, Directed Imagery Technique (DIT), is an effective, economical and therapeutic technique that can be easily used in nursing practices. YIT is a set of stories that individuals create by visualizing the symbols given by the practitioner after relaxation exercises. Within the scope of this technique, which is a window to the inner world of the person, the creation of one's own unique story through symbols is encouraged. This randomized controlled experimental study will be conducted to evaluate the effect of guided imagery supported psychoeducation on depression, self-esteem and stress levels of individuals diagnosed with depression. The population of the study will consist of individuals diagnosed with depression who applied to Kilis Alaeddin Yavaşça State Hospital Psychiatry Outpatient Clinic. The sample of the study will consist of 60 individuals (30 experimental and 30 control) who applied to Kilis Alaeddin Yavaşça State Hospital Psychiatry Outpatient Clinic and agreed to participate in the study. In both groups, a face-to-face interview technique will be used to administer the Introductory Information Form, Beck Depression Scale (BDS), Rosenberg Self-Esteem Scale (RBSS) and Perceived Stress Scale (PSS) and the responses of the individuals will be recorded. The experimental group will be administered individually face-to-face twice a week for a total of three weeks. In addition, the audio recording made in a professional studio environment will be used for individuals to listen at home. Individuals will be instructed to listen to the audio recording twice a week for three weeks starting from the second week when the researcher started to apply the imagery technique. After the interventions applied to the experimental group are over, the scales will be applied again to the individuals in the experimental and control groups.

DETAILED DESCRIPTION:
PROBLEM STATEMENT Depressive disorder is a common mental disorder. Its classic symptoms include depressed mood, anxiety, anhedonia, and cognitive impairments that deeply affect quality of life. Depression is one of the leading causes of disability worldwide and is a primary cause of deaths by suicide. Approximately 5% of adults globally (4% in men and 6% in women), including 5.7% of those aged 60 and older, suffer from depression, accounting for 3.8% of the total population. It is estimated that around 280 million people worldwide have depression.

Depression is often referred to as a disorder related to stress, and it is known that stress caused by negative life events, including early life experiences, contributes to the onset, development, and progression of this disorder. Studies indicate that high levels of exposure to negative stressors significantly contribute to cases of depression, emphasizing the importance of timely recognition of stress exposure in these individuals.

Research has also revealed that self-esteem plays a significant role in depression. Self-esteem is defined as "a person's specific attitude and perception regarding themselves and their interactions with others" . Low self-esteem has been empirically shown to be a risk factor for the development of depression and suicidal thoughts. Low self-esteem is a symptom of depressive disorders and is considered by some as a precursor to relapse, while high self-esteem seems to act as a buffer against depression.

Despite the availability of effective treatments for depression, not all patients receive treatment, and a significant portion of those who do do not recover. There is an increasing need for low-cost and easily accessible new methods to cope with the health burden created by depression. There are various psychological interventions for treating depression, and one of the effective ones is psychoeducation. Psychoeducational programs are designed to help individuals with mental disorders understand and manage their conditions. This is achieved by empowering patients' resources and skills so they can cope better with their situations, prevent relapses, and contribute to their health and well-being. Studies have indicated that psychoeducational programs have positive effects on depression.

Another method, Guided Imagery Technique (GIT), is an effective, economical, and therapeutic technique that can be easily used in nursing practices. GIT consists of a series of stories created by individuals through visualizing symbols given by the practitioner after relaxation exercises. This technique, which opens a window to the individual's inner world, encourages the creation of their unique story through symbols. It has been shown that this technique positively affects vital signs, electroencephalography patterns, blood flow, gastric motility and secretions, sexual arousal, and various hormone and neurotransmitter levels. Guided imagery has been found to reduce depression, anxiety, stress, pain, and chemotherapy-related side effects, increase empathy levels, decrease symptoms of post-traumatic stress disorder, lower high blood pressure, enhance quality of life, and strengthen the immune system. It is noted that the application of guided imagery techniques in psychiatric patients is limited in national and international literature.

This research aims to determine the effects of guided imagery-supported psychoeducation on depression, self-esteem, and stress levels in individuals diagnosed with depression, which is expected to raise awareness both individually and socially regarding the disease of depression, and the identified risk factors will guide interventions. Additionally, the research is anticipated to serve as a guide for psychiatric nurses and community mental health nurses in applying guided imagery techniques and for future studies related to guided imagery in psychiatric disorders.

Research Hypotheses H0 Hypothesis: Guided imagery-supported psychoeducation applied to individuals diagnosed with depression does not affect the depression, self-esteem, and stress levels of patients in the experimental and control groups.

H1a Hypothesis: Guided imagery-supported psychoeducation applied to individuals diagnosed with depression will result in a decrease in the average depression scores of patients in the experimental group compared to those in the control group.

H1b Hypothesis: Guided imagery-supported psychoeducation applied to individuals diagnosed with depression will lead to an increase in the average self-esteem scores of patients in the experimental group compared to those in the control group.

H1c Hypothesis: Guided imagery-supported psychoeducation applied to individuals diagnosed with depression will result in a decrease in the average stress scores of patients in the experimental group compared to those in the control group.

H2 Hypothesis: Guided imagery-supported psychoeducation applied to individuals diagnosed with depression will lead to a decrease in the average depression and stress scores of patients in the experimental group after the intervention compared to before, while increasing their average self-esteem scores.

MATERIALS AND METHODS Research Type This research is a randomized controlled experimental study.

Research Population and Sample The population of the study will consist of individuals diagnosed with depression who apply to the Psychiatry Clinic of Kilis Alaeddin Yavaşça State Hospital and meet the inclusion criteria for the study. The sample size will be calculated using the G-Power program. The experimental and control groups will be determined based on randomization.

The sample selection criteria for the study are expressed in Table 1.

Table 1: Sample Selection Criteria of the Study

Inclusion Criteria Exclusion Criteria

* Be 18 years of age or older • Be under 18 years of age
* Be literate • Be illiterate
* Be followed for at least one month with a diagnosis of depression according to DSM V criteria and receiving medication treatment • Not being followed with a diagnosis of depression according to DSM V criteria and not receiving medication treatment
* No history of suicide attempts • History of suicide attempts
* Not having received ECT in the last year • Having received ECT in the last year
* No cognitive and communication barriers that would prevent them from sustaining the interview and completing the questionnaires • Having comorbid mental illness
* Be able to use a smartphone • Not agreeing to participate after information
* Agree to participate after being informed Data Collection and Research Process The research will be conducted between May 2024 and May 2025 at the Psychiatry Clinic of Kilis Alaeddin Yavaşça State Hospital. The data collection tools will include an Introductory Information Form, Beck Depression Inventory (BDI), Rosenberg Self-Esteem Scale (RSES), and Perceived Stress Scale (PSS).

Individuals in the experimental and control groups will be interviewed separately to provide information about the study and obtain their written consent. After applying the introductory information form and scales, guided imagery-supported psychoeducation will be applied to the experimental group. After the study is completed, the guided imagery-supported psychoeducation program will also be applied to the control group.

Application of Guided Imagery-Supported Psychoeducation The guided imagery-supported psychoeducation to be applied to the experimental group will be created with expert consultation. The researcher has received training in Guided Imagery Technique.

Guided imagery-supported psychoeducation will be applied to the experimental group face-to-face twice a week for a total of three weeks to reduce depression levels, increase self-esteem, and decrease perceived stress levels. Additionally, a professionally recorded audio will be provided for individuals to listen to at home. Participants will be instructed to listen to the audio recording twice a week for three weeks starting from the second week when the researcher begins applying the imagery technique. Literature indicates that the duration of GIT applied to individuals with depression varies between a total of 8 to 12 sessions. Therefore, the study is planned to consist of a total of 14 sessions.

Sessions will begin with an introduction and the application of scales. The first two sessions will consist of a psychoeducation program containing information about depressive disorders, self-esteem, perceived stress, the relationship between these concepts, and the guided imagery technique. In subsequent sessions, the Guided Imagery Technique will be applied. The application will include relaxation exercises, the imagery process, and steps for relaxation. During the imagery process, participants will be asked to close their eyes. The metaphors of meadow, stream, and house will be used. The meadow metaphor is preferred at the beginning of the imagery as it allows the individual to feel safe. The stream metaphor will then symbolize the flow of life. The house metaphor is thought to symbolize the individual's personality. It is expressed that the house metaphor is related to self-esteem in GIT. After the house metaphor, positive imagery will be conducted to enhance self-esteem and alleviate stress, followed by a body-oriented relaxation and return to the main focus to conclude the application.

During the initial interview when pre-tests are conducted, participants will be informed about the important points to consider. Before the application, participants will be instructed to listen to the audio recording at the most suitable time of the day for them, in a place where they will not be disturbed by others, and to put their phones on airplane mode while using headphones. During the interview, the script of the scenario will be read to the participants, and any unclear points will be explained. Participants will be informed that they will receive a reminder call to ensure they listen to the audio recordings and their consent will be obtained. Participants who listen to the audio recordings will be asked to note the date and time of each listening, as well as what they felt and thought after listening. During the first interview, the audio recordings will be transferred to the participants' phones via computer. After the interventions applied to the experimental group are completed, the scales will be reapplied to both the experimental and control groups.

Data Collection Tools Introductory Information Form: This form, prepared by the researcher, contains the sociodemographic characteristics of the participants and information related to the disease, consisting of 19 questions.

Beck Depression Inventory (BDI): Developed by Beck and colleagues in 1961 to measure somatic, emotional, cognitive, and motivational symptoms seen in depression. The Turkish validity and reliability study of the scale was conducted by Hisli in 1988. The scale has four response options [a (0), b (1), c (2), d (3) points] and consists of 21 items. The highest score that can be obtained from the scale is 63. A higher total score indicates a higher level or severity of depression. According to the total score, the severity of depression is interpreted as "0-9=Minimal, 10-16=Mild, 17-29=Moderate, 30-63=Severe." The reliability coefficient of the Turkish form of the scale was determined to be 0.80.

Rosenberg Self-Esteem Scale (RSES): Developed by Rosenberg in 1965 to measure individuals' self-esteem. The Turkish validity and reliability study of the scale was conducted by Çuhadaroğlu in 1986. The self-esteem subtest of the scale consists of 10 items. The highest score that can be obtained from the scale is 6, and lower scores indicate higher self-esteem. Those scoring 0-1 are considered to have high self-esteem, 2-4 medium self-esteem, and 5-6 low self-esteem. The reliability coefficient of the Turkish form of the scale was determined to be 0.71.

Perceived Stress Scale (PSS): Developed by Cohen, Kamarck, and Mermelstein in 1983 to determine how stressful individuals perceive certain situations in their lives. The Turkish validity and reliability study of the scale was conducted by Eskin et al. in 2013. The items in the scale are answered on a five-point Likert scale ranging from "Never (0)" to "Very Often (4)" and consist of a total of 14 items. Seven items (items 4, 5, 6, 7, 9, 10, 13) are reverse scored. The scale has two subscales: self-efficacy and stress perception. The lowest score that can be obtained from the scale is 0, and the highest score is 56. Higher scores indicate a higher perception of stress. The reliability coefficient of the Turkish form of the scale was determined to be 0.84.

Statistical Analysis of Data Statistical analyses of the research will be conducted using the SPSS 22 software. The normal distribution of the data will be evaluated using the Shapiro-Wilk test, Kolmogorov-Smirnov tests, skewness, and kurtosis values. Parametric tests will be used to evaluate data that conform to normal distribution. In the evaluation of the data, descriptive statistics such as percentage, arithmetic mean, and standard deviation will be used for the distribution of the descriptive characteristics of the patients in the experimental and control groups. The descriptive statistics of the total scale scores of the patients in the experimental and control groups will include mean and standard deviation; independent samples t-test will be used to compare the pre-test scale score means of the patients in the experimental and control groups; independent samples t-test will be used to compare the post-test scale score means of the patients in the experimental and control groups; variance analysis will be used for within-group comparisons of the pre-post test scale score means of the experimental group; and variance analysis will be used for within-group comparisons of the pre-post test scale score means of the control group. In all analyses, a confidence interval of 95% and a significance level of p<0.05 will be accepted.

Dependent and Independent Variables of the Research Dependent Variables: Average scores of Beck Depression Inventory, average scores of Rosenberg Self-Esteem Scale, average scores of Perceived Stress Scale.

Independent Variable: Guided imagery-supported psychoeducation. Ethical Aspects of the Research Approval from the Clinical Research Ethics Committee of Kilis 7 December University will be obtained to conduct the research. Additionally, written permission will be obtained from the Kilis Provincial Health Directorate.

Participants will be informed about the purpose of the research and the content of the forms, and verbal consent will be obtained from them, followed by signing the "Informed Consent Form." Questions that participants do not understand or wish to ask about the research will be answered. Participants will be informed that they are free to participate in the research voluntarily without any pressure and can withdraw from the research at any time, respecting the principle of "Respect for Autonomy," and that their information will remain confidential, adhering to the principle of "Confidentiality and Protection of Privacy."

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* To be literate
* Being followed up with a diagnosis of depression according to DSM V criteria for at least one month and receiving medication
* Not being a suicide attempt
* Not having received ECT in the last 1 year
* No cognitive and communication disabilities that would prevent continuing the interview and completing the questionnaires
* Being able to use a smartphone
* To agree to participate in the study after being informed

Exclusion Criteria:

* - Under 18 years of age
* Illiteracy
* Not being followed up with a diagnosis of depression according to DSM V criteria for at least one month and not receiving medication
* Being a suicide attempt
* Having received ECT within the last 1 year
* Comorbid mental illness
* Having cognitive and communication disabilities that would prevent continuing the interview and completing the questionnaires
* Refusing to participate in the study after being informed

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-12-23 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Depression level | Day 1
  The level of depression will be measured with the Beck Depression Scale. The level of depression severity is interpreted as "0-9=minimal, 10-16=mild, 17-29=moderate, 30-63=severe" according to the total score.
Self-esteem | Day 1
  Self-esteem level will be measured with the Rosenberg Self-Esteem Scale. Those who score 0-1 on the scale are considered to have high self-esteem, those who score 2-4 are considered to have medium self-esteem, and those who score 5-6 are considered to have low self-esteem.
Stress | Day 1
  The stress level will be measured with the Perceived Stress Scale. The lowest score that can be obtained from the scale is 0, the highest score is 56. High scores obtained from the scale indicate that the individual's perception of stress is high.
Stress | up to four weeks
  The stress level will be measured with the Perceived Stress Scale. The lowest score that can be obtained from the scale is 0, the highest score is 56. High scores obtained from the scale indicate that the individual's perception of stress is high.

SECONDARY OUTCOMES:
Depression level | up to four weeks
  The level of depression will be measured with the Beck Depression Scale. The level of depression severity is interpreted as "0-9=minimal, 10-16=mild, 17-29=moderate, 30-63=severe" according to the total score.
Self-esteem | up to four weeks
  Self-esteem level will be measured with the Rosenberg Self-Esteem Scale. Those who score 0-1 on the scale are considered to have high self-esteem, those who score 2-4 are considered to have medium self-esteem, and those who score 5-6 are considered to have low self-esteem.

CONTACTS AND LOCATIONS:
Locations (1):
- Kilis 7 Aralik University, Kilis, Turkey (Türkiye)